CLINICAL TRIAL: NCT03410225
Title: Computer-Assisted Motivational Interviewing Intervention to Facilitate Teen Pregnancy Prevention and Fitness Behavior Changes: A Randomized Trial for Young Men
Brief Title: Motivational Interviewing for Getting Healthy TodaY Study
Acronym: MIGHTY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: The Office of Adolescent Health, HHS (U.S. Federal Agency); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAR5303
Record Dates: First submitted 2018-01-09; First posted 2018-01-25 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Pregnancy Related; Diet Modification
Keywords: Pregnancy Prevention; Male Involvement
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be randomized through a permuted random blocks assignment procedure with block stratification (by age group). Strings of varying length (2, 4, 6, 8, for example), with equal allocations T and C (randomly ordered) within a string, are combined to produce a single, long string of T and C combinations (e.g. TTCCTCTTCCC, etc.). Because the long string is made up of blocks of T and C strings with equal allocations of Ts and Cs, the observed percentage of the sample in the treatment condition will always be very close to 0.5, and the true P(T) for all observations will be 0.5. Randomization will be conducted via an algorithm on the online portal at the time of enrollment in order for the project coordinator to assign the participant to an intervention arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAMI-TPP (Experimental): Young men, ages 15 to 24 years, will be receiving a modified CAMI aimed at Teen Pregnancy Prevention (CAMI-TPP).
  Interventions: Behavioral: CAMI-TPP
- CAMI-Fitness (Active Comparator): Young men, ages 15 to 24 years, will be receiving CAMI aimed at healthy diet, physical activity and tobacco avoidance (CAMI-Fitness).
  Interventions: Behavioral: CAMI-Fitness

INTERVENTIONS:
Behavioral: CAMI-TPP — The TPP group will receive four 30-minute sessions of one-on-one coaching over 12 weeks with a MI coach; the sessions will be guided by personalized feedback aimed at increasing condom use, supporting female partners in contraceptive use, and obtaining reproductive health services and STI testing. MI counseling sessions will be conducted by phone or video call.
  Other Names: CAMI - Teen Pregnancy Prevention
  Arms: CAMI-TPP
Behavioral: CAMI-Fitness — The Fitness group will also receive four 30-minute sessions of one-on-one coaching over 12 weeks with a MI coach; these sessions will be guided by personalized feedback aimed at healthy diet, physical activity and tobacco avoidance. MI counseling sessions will be conducted by phone or video call.
  Other Names: CAMI - healthy diet, physical activity and tobacco avoidance
  Arms: CAMI-Fitness

SUMMARY:
The present study aims to test and rigorously evaluate the effectiveness of a computer-assisted motivational interviewing (CAMI) intervention that has already been shown to be successful with young women by reducing the risk of rapid subsequent birth among adolescent mothers, and applying this intervention to young men.

The purpose of the intervention is to increase condom use, increase female partner use of moderately or highly effective contraception, and increase completion of a reproductive health visit and STI/HIV testing.

The primary hypothesis is that the CAMI-TPP (CAMI aimed at Teen Pregnancy Prevention) intervention will increase the proportion of participants who do not engage in risky sex, report condom use at last intercourse as well as partner use of contraception compared to those in the Fitness group. It is also predicted that young men who receive the CAMI-TPP will report higher completion of a reproductive health service visit with sexually transmitted infection (STI) testing over the course of study participation compared to those in the CAMI-Fitness (CAMI aimed at healthy diet, physical activity and tobacco avoidance) group.

DETAILED DESCRIPTION:
Most teen pregnancies (82%) in the United States are unintended. Actively engaging young men in preventing teen pregnancy is a necessary and central component to effecting change. Young men, aged 15-19 and 20-24 years, father most of the children born to teen mothers. Few interventions have been designed specifically or shown to be effective for young men in reducing teen pregnancy.

Counseling and feedback based on Motivational Interviewing (MI) principles demonstrated greater success than standard, didactic advice in several domains of behavior change. The effectiveness of this type of counseling to alter young men's sexual and contraceptive behaviors has not been rigorously evaluated.

Participants will be randomly chosen (like flipping a coin) to take part in one of the two MI projects, and you will get coaching and use an app for that project to improve your health. One project is on teen pregnancy prevention and the other is on healthy eating, physical activity, and avoiding cigarettes. Participants will use an app via phone to do the project, answer survey questions, keep track of health, and learn more about healthy behaviors.

Three hundred young men, ages 15 to 24 years, will be randomized to one of two intervention arms, a modified CAMI aimed at Teen Pregnancy Prevention (CAMI-TPP) or a CAMI aimed at healthy diet, physical activity and tobacco avoidance (CAMI-Fitness). The two interventions are identical in length and timing but vary in the target behavior focus (pregnancy prevention versus fitness).

ELIGIBILITY:
Inclusion Criteria:

* Young men aged 15-24
* Sexually active with female partners
* Enrolled patients at New York Presbyterian Hospital's Young Men's Clinic (YMC) in Washington Heights or the school-based health centers (SBHCs) at George Washington Educational Campus in Washington Heights or John F. Kennedy campus in the Bronx

Exclusion Criteria:

* Do not have iPhone or Android Smartphone
* Participated in any of the following programs within the last year, or have a brother who has participated in these programs:

  * Fathers Raising Responsible Men (FRRM)
  * Peer Group Connection (PGC)
  * NYC Teens Connection
  * Children's AID Society (CAS)-TPP Initiative
  * Achieving Condom Empowerment-Plus (ACE+) Study
* Have had a medical treatment or surgical procedure that makes it impossible to father a child, such as a vasectomy
* Cannot commit to participating in a smartphone-based study for the next 15 months

Ages: 15 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Change in number of participants that had sexual intercourse without using a condom since the last assessment Condom use at last sex | Baseline and 12 weeks
  In the past 3 months, how many times have you had sexual intercourse without using a condom?

SECONDARY OUTCOMES:
Change in number of participants that had sexual intercourse in the past without the partner using any contraception since the last assessment | Baseline and 12 weeks
  In the past 3 months, how many times have you had sexual intercourse without using any of these methods of birth control?
Number of participants completing a reproductive health service visit with STI testing | Baseline and 12 weeks
  In the last 3 months, that is, since {current date minus 3 months} , have you been tested by a doctor, nurse, or health provider for a sexually transmitted disease like gonorrhea, chlamydia, herpes, or syphilis (not including HIV)?

CONTACTS AND LOCATIONS:
Overall Officials: David L. Bell, MD, MPH, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - George Washington Educational Campus School-Based Health Center, New York, New York
  - The Young Men's Clinic, New York, New York
  - John F. Kennedy Educational Campus School-Based Health Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finer LB, Zolna MR. Shifts in intended and unintended pregnancies in the United States, 2001-2008. Am J Public Health. 2014 Feb;104 Suppl 1(Suppl 1):S43-8. doi: 10.2105/AJPH.2013.301416. Epub 2013 Dec 19. PMID 24354819
- [Background] Martin JA, Hamilton BE, Ventura SJ, Osterman MJ, Wilson EC, Mathews TJ. Births: final data for 2010. Natl Vital Stat Rep. 2012 Aug 28;61(1):1-72. PMID 24974589
- [Background] Males MA. Adult involvement in teenage childbearing and STD. Lancet. 1995 Jul 8;346(8967):64-5. doi: 10.1016/s0140-6736(95)92105-2. PMID 7603210
- [Background] Hollis JF, Polen MR, Whitlock EP, Lichtenstein E, Mullooly JP, Velicer WF, Redding CA. Teen reach: outcomes from a randomized, controlled trial of a tobacco reduction program for teens seen in primary medical care. Pediatrics. 2005 Apr;115(4):981-9. doi: 10.1542/peds.2004-0981. PMID 15805374
- [Background] McCambridge J, Strang J. The efficacy of single-session motivational interviewing in reducing drug consumption and perceptions of drug-related risk and harm among young people: results from a multi-site cluster randomized trial. Addiction. 2004 Jan;99(1):39-52. doi: 10.1111/j.1360-0443.2004.00564.x. PMID 14678061
- [Background] Weinstein P, Harrison R, Benton T. Motivating mothers to prevent caries: confirming the beneficial effect of counseling. J Am Dent Assoc. 2006 Jun;137(6):789-93. doi: 10.14219/jada.archive.2006.0291. PMID 16803808
- [Background] Jensen CD, Cushing CC, Aylward BS, Craig JT, Sorell DM, Steele RG. Effectiveness of motivational interviewing interventions for adolescent substance use behavior change: a meta-analytic review. J Consult Clin Psychol. 2011 Aug;79(4):433-40. doi: 10.1037/a0023992. PMID 21728400
- [Background] Channon SJ, Huws-Thomas MV, Rollnick S, Hood K, Cannings-John RL, Rogers C, Gregory JW. A multicenter randomized controlled trial of motivational interviewing in teenagers with diabetes. Diabetes Care. 2007 Jun;30(6):1390-5. doi: 10.2337/dc06-2260. Epub 2007 Mar 10. PMID 17351283